CLINICAL TRIAL: NCT02972138
Title: Vitamin D Supplementation and Anti-resorptive Therapy (Bisphosphonates) Treatment of Young Adult Patients With Sickle Cell Disease
Brief Title: Vitamin D and Bisphosphonates in the Treatment of Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Responsible Party: Sponsor
Other Study IDs: Vit.D-Bisph-SCD
Record Dates: First submitted 2016-10-28; First posted 2016-11-23 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-12

CONDITIONS: Sickle Cells Disease
Keywords: Sickle-cells Disease; bisphosphonates; Vitamine D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sickle cell disease (SCD) is a worldwide distributed hereditary red cell disorder, which affects approximately 75,000 individuals in the United States and almost 20,000- 25,000 subjects in Europe, this latter mainly related to the immigration fluxes from endemic areas such as Sub-Saharian Africa to European countries. Studies of global burden disease have pointed out the invalidating impact of SCD on patient quality of life. This requires the development of new therapeutic options to treat sickle cell related acute and chronic complications. SCD is caused by a point mutation in the β-globin gene resulting in the synthesis of pathological hemoglobin S (HbS). HbS displays peculiar biochemical characteristics, polymerizing when deoxygenated with associated reduction in cell ion and water content (cell dehydration), increased red cell density and further acceleration of HbS polymerization. Pathophysiological studies have shown that dense, dehydrated red cells play a central role in acute and chronic clinical manifestations of SCD, in which intravascular sickling in capillaries and small vessels leads to vaso-occlusion and impaired blood flow with ischemic/reperfusion injury. In microcirculation, vaso-occlusive events (VOC) result from a complex and still partially known scenario, involving the interactions between different cell types, including dense red cells, reticulocytes, abnormally activated endothelial cells, leukocytes, platelets and plasma factors. Target organs, such as bone or lung, are involved in both acute and chronic clinical manifestations of SCD, related to their peculiar anatomic organization mainly characterized by sluggish circulation and relative local hypoxia. VOCs combined with marrow hyperplasia and inflammation has been suggested to contribute to the development of sickle bone disease (SBD). Recently, it has been proposed a possible role of vitamin D deficiency in SBD, which appears to be subordinated to the primary defect in bone homeostasis. In a humanized mouse model for SCD, we recently reported that SBD is due to imbalance between osteoblast/osteoclast activity induced by recurrent VOCs. In addition, we show that zoledronic acid prevents bone impairment related to SCD, reducing osteoclast activity and improving osteoblast performance.

DETAILED DESCRIPTION:
This is a retrospective study aimed to evaluate sickle bone disease (SBD) in a population of young adult patients with sickle cell disease treated with vitamin D supplementation and anti-resorptive therapy (bisphosphonates). We plan to analyze data from 1 January 2010 to 31 December 2015.

In addition to the standard hematological analysis, the following parameters and radiologic exams will be evaluated:

* Serum levels of Ca2+, P, Vitamin D, parathormone , creatinine, blood urea nitrogen , Na, K, Cl
* Bone turnover markers: C-terminal telopeptide (CTX), N-terminal propeptide of type I procollagen (PINP)
* Bone densitometry (DXA) at lumbar spine and proximal femur
* Standard X-Ray at dorsal-lumbar spine in LL projection for morphometric analysis

ELIGIBILITY:
Inclusion Criteria:

* Young adult patients with sickle cell disease (older than 18 years of age) and younger than 50 years of age

Exclusion Criteria:

* Women with positive pregnant test, patients with history of heart, renal and liver failure, patients taking drugs influencing bone metabolisms within the two years before the beginning of the study (i.e.: glucocorticoids, hormonal replacement)
* Patients in meonopause, patients with traumatic vertebral fracture
* Patients with hypo/hyperthyroidism
* Patients with hyperparathyroidism
* Patients with osteomalacia, patients with history of Paget disease
* Patients with Cushing syndrome
* Patients with malabsorption diseases (i.e.: caeliac disease)
* Patients with history of cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with sickle cell disease older than 18 years of age and younger than 50 years of age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence of vertebral fracture | 5 years follow up

SECONDARY OUTCOMES:
severity of vertebral fracture | 5 years follow up
Incidence of non-vertebral fracture | 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Luca G Dalle Carbonare, MD, Principal Investigator — Università degli studi di Verona
Locations (3):
- Italy (3):
  - Ospedali Galliera - S.S.D. Microcitemia, anemie congenite e dismetabolismo del ferro, Genova
  - Ospedali Galliera - S.S.D. Ortogeriatria per intensità di cure, Genova
  - Università degli Studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Modell B, Darlison M. Global epidemiology of haemoglobin disorders and derived service indicators. Bull World Health Organ. 2008 Jun;86(6):480-7. doi: 10.2471/blt.06.036673. PMID 18568278
- [Background] Weatherall DJ, Clegg JB. Inherited haemoglobin disorders: an increasing global health problem. Bull World Health Organ. 2001;79(8):704-12. Epub 2001 Oct 24. PMID 11545326
- [Background] De Franceschi L, Cappellini MD, Olivieri O. Thrombosis and sickle cell disease. Semin Thromb Hemost. 2011 Apr;37(3):226-36. doi: 10.1055/s-0031-1273087. Epub 2011 Mar 31. PMID 21455857
- [Background] Eaton WA, Hofrichter J. Sickle cell hemoglobin polymerization. Adv Protein Chem. 1990;40:63-279. doi: 10.1016/s0065-3233(08)60287-9. No abstract available. PMID 2195851
- [Background] De Franceschi L, Corrocher R. Established and experimental treatments for sickle cell disease. Haematologica. 2004 Mar;89(3):348-56. PMID 15020275
- [Background] Ballas SK, Smith ED. Red blood cell changes during the evolution of the sickle cell painful crisis. Blood. 1992 Apr 15;79(8):2154-63. PMID 1562742
- [Background] Vinchi F, De Franceschi L, Ghigo A, Townes T, Cimino J, Silengo L, Hirsch E, Altruda F, Tolosano E. Hemopexin therapy improves cardiovascular function by preventing heme-induced endothelial toxicity in mouse models of hemolytic diseases. Circulation. 2013 Mar 26;127(12):1317-29. doi: 10.1161/CIRCULATIONAHA.112.130179. Epub 2013 Feb 27. PMID 23446829
- [Background] Hebbel RP, Vercellotti G, Nath KA. A systems biology consideration of the vasculopathy of sickle cell anemia: the need for multi-modality chemo-prophylaxsis. Cardiovasc Hematol Disord Drug Targets. 2009 Dec;9(4):271-92. doi: 10.2174/1871529x10909040271. PMID 19751187
- [Background] Hebbel RP. Adhesion of sickle red cells to endothelium: myths and future directions. Transfus Clin Biol. 2008 Feb-Mar;15(1-2):14-8. doi: 10.1016/j.tracli.2008.03.011. Epub 2008 May 23. PMID 18501652
- [Background] Platt OS. The acute chest syndrome of sickle cell disease. N Engl J Med. 2000 Jun 22;342(25):1904-7. doi: 10.1056/NEJM200006223422510. No abstract available. PMID 10861328
- [Background] Lal A, Fung EB, Pakbaz Z, Hackney-Stephens E, Vichinsky EP. Bone mineral density in children with sickle cell anemia. Pediatr Blood Cancer. 2006 Dec;47(7):901-6. doi: 10.1002/pbc.20681. PMID 16317761
- [Background] Dalle Carbonare L, Innamorati G, Valenti MT. Transcription factor Runx2 and its application to bone tissue engineering. Stem Cell Rev Rep. 2012 Sep;8(3):891-7. doi: 10.1007/s12015-011-9337-4. PMID 22139789
- [Background] Bruzzaniti A, Baron R. Molecular regulation of osteoclast activity. Rev Endocr Metab Disord. 2006 Jun;7(1-2):123-39. doi: 10.1007/s11154-006-9009-x. PMID 16951988
- [Background] Dalle Carbonare L, Zanatta M, Gasparetto A, Valenti MT. Safety and tolerability of zoledronic acid and other bisphosphonates in osteoporosis management. Drug Healthc Patient Saf. 2010;2:121-37. doi: 10.2147/DHPS.S6285. Epub 2010 Aug 19. PMID 21701624
- [Background] Dalle Carbonare L, Arlot ME, Chavassieux PM, Roux JP, Portero NR, Meunier PJ. Comparison of trabecular bone microarchitecture and remodeling in glucocorticoid-induced and postmenopausal osteoporosis. J Bone Miner Res. 2001 Jan;16(1):97-103. doi: 10.1359/jbmr.2001.16.1.97. PMID 11149495
- [Background] Nouraie M, Cheng K, Niu X, Moore-King E, Fadojutimi-Akinsi MF, Minniti CP, Sable C, Rana S, Dham N, Campbell A, Ensing G, Kato GJ, Gladwin MT, Castro OL, Gordeuk VR. Predictors of osteoclast activity in patients with sickle cell disease. Haematologica. 2011 Aug;96(8):1092-8. doi: 10.3324/haematol.2011.042499. Epub 2011 May 5. PMID 21546502
- [Background] Neves FS, Oliveira LS, Torres MG, Toralles MB, da Silva MC, Campos MI, Campos PS, Crusoe-Rebello I. Evaluation of panoramic radiomorphometric indices related to low bone density in sickle cell disease. Osteoporos Int. 2012 Jul;23(7):2037-42. doi: 10.1007/s00198-011-1810-z. Epub 2011 Oct 18. PMID 22006042
- [Background] Nur E, Mairuhu W, Biemond BJ, van Zanten AP, Schnog JJ, Brandjes DP, Otten HM; CURAMA study group. Urinary markers of bone resorption, pyridinoline and deoxypyridinoline, are increased in sickle cell patients with further increments during painful crisis. Am J Hematol. 2010 Nov;85(11):902-4. doi: 10.1002/ajh.21856. PMID 20882525
- [Background] Miller RG, Segal JB, Ashar BH, Leung S, Ahmed S, Siddique S, Rice T, Lanzkron S. High prevalence and correlates of low bone mineral density in young adults with sickle cell disease. Am J Hematol. 2006 Apr;81(4):236-41. doi: 10.1002/ajh.20541. PMID 16550513